CLINICAL TRIAL: NCT05440760
Title: Using Virtual Reality Technology to Improve Patient Experience and Quality of Care During Brachytherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 261231
Record Dates: First submitted 2022-06-20; First posted 2022-07-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Endocervical Cancer
Keywords: Brachytherapy; Virtual Reality

STUDY DESIGN:
Intervention Model Description: Subjects will be placed into four treatment-sequence groups in a 1:1:1:1 allocation ratio via permuted block randomization with randomized block sizes of four or eight.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sequence Group A (Experimental): VR distraction occurring visits 1 and 2 with normal SOC therapy at visits 3 and 4.
  Interventions: Device: The Oculus Quest 2 Virtual Reality Headset
- Sequence Group B (Experimental): VR distraction occurring visits 1 and 4 with normal SOC therapy at visits 2 and 3.
  Interventions: Device: The Oculus Quest 2 Virtual Reality Headset
- Sequence Group C (Experimental): VR distraction occurring visits 3 and 4 with normal SOC therapy at visits 1 and 2.
  Interventions: Device: The Oculus Quest 2 Virtual Reality Headset
- Sequence Group D (Experimental): VR distraction occurring visits 2 and 3 with normal SOC therapy at visits 3 and 4.
  Interventions: Device: The Oculus Quest 2 Virtual Reality Headset

INTERVENTIONS:
Device: The Oculus Quest 2 Virtual Reality Headset — The hardware includes the wireless headset with integrated headphones which will block the sight and sounds of the clinical setting as well as the hand controllers for the interactive VR experience, which will be delivered through any of three VR software options (subject may choose one or more from the following options):
  * Titans of Space® PLUS developed by Drash VR, LLC (Murrieta, CA, USA)
  * TRIPP® developed by TRIPP, Inc. (Los Angeles, CA, USA)
  * Nature Treks VR published by Greener Games (Ironbridge, England, UK)

SUMMARY:
The primary objective is to demonstrate the feasibility of incorporating VR distraction into the brachytherapy and radiotherapy clinical workflow.

The secondary objective is to determine if VR distraction during brachytherapy treatment for cervical cancer improves subjects' satisfaction, procedural/acute pain, and need for analgesics or anxiolytics.

DETAILED DESCRIPTION:
This will be a prospective pilot study conducted at UAMS. All subjects will experience VR distraction using a crossover design in which each subject receives four rounds of brachytherapy: two rounds with VR distraction and two rounds without VR distraction. Brachytherapy will be conducted per SoC workflow. Subjects will be placed into four treatment-sequence groups in a 1:1:1:1 allocation ratio via permuted block randomization with randomized block sizes of four or eight.

The four treatment-sequence groups will follow the four-session treatment schedules outlined below, in which "V" denotes the sessions when VR distraction is used while "N" denotes the sessions when it is not:

* Sequence Group A will be treated according to schedule VVNN.
* Sequence Group B will be treated according to schedule VNNV.
* Sequence Group C will be treated according to schedule NNVV.
* Sequence Group D will be treated according to schedule NVVN.

ELIGIBILITY:
Inclusion Criteria:

* Female, ≥ 18 years of age
* Histopathologic diagnosis of gynecologic cancer (endometrial, cervical, vaginal, vulvar) that requires intracavitary brachytherapy with a tandem or interstitial brachytherapy
* Able to provide written consent

Exclusion Criteria:

* Severe vision or hearing problems that may hinder the ability to see or hear clearly through the VR headset or other condition that may interfere with the placement of the VR headset such as a head, ear or facial wound
* History of seizure disorder, severe motion sickness, dizziness, or migraine headaches precipitated by visual auras
* Known history of elevated intraocular pressure
* Claustrophobia, thalassophobia, cleithrophobia or similar phobias
* Any other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment regimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The number of eligible subjects who enroll onto the study. | 3 weeks
The number of subjects who withdraw or are withdrawn from the study. | 3 weeks
The number of subjects who successfully complete the study questionnaires for satisfaction, procedural pain, and anxiety. | 3 weeks
The number of times a technical problem occurs with the VR distraction | 3 weeks

SECONDARY OUTCOMES:
Determination of VR distraction during brachytherapy treatment for cervical cancer pain | 3 weeks
  Compare the subject's procedural pain scores (using a visual analog scale [VAS] pre- and post-procedure) between sessions with VR and sessions without VR.
Determination of VR distraction during brachytherapy treatment for cervical cancer on anxiety. | 3 weeks
  Compare the subject's procedural anxiety scores (using a VAS pre- and post-procedure) between sessions with VR and sessions without VR.
Opiod dose | 3 weeks
  Compare the dose(s) of opioid pain medication per session (using morphine milligram equivalents [MMEs]) between sessions with VR and sessions without VR.
Benzodiazepine dose | 3 weeks
  Compare the dose(s) of benzodiazepine anxiolytics per session (using a benzodiazepine conversion calculator) between sessions with VR and sessions without VR

CONTACTS AND LOCATIONS:
Overall Officials: Gary Lewis, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States